CLINICAL TRIAL: NCT01946412
Title: A Phase 3, 2-Arm, Roll-Over Study to Evaluate the Long-term Safety and Pharmacodynamics of Ivacaftor Treatment in Pediatric Subjects With Cystic Fibrosis and a CFTR Gating Mutation
Brief Title: Roll-Over Study of Ivacaftor in Cystic Fibrosis Pediatric Subjects With a CF Transmembrane Conductance Regulator Gene (CFTR) Gating Mutation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VX11-770-109
Record Dates: First submitted 2013-09-16; First posted 2013-09-19 (Estimated); Results first posted 2017-02-01 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2016-12

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — ivacaftor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Observational Arm (No Intervention)
- Ivacaftor (Experimental): Ivacaftor will be administered every 12 hours (q12h) from Day 1 through the Week 84 Visit. The ivacaftor dose will be:
  * 50 mg q12h for subjects 2 to <6 years of age and <14 kg,
  * 75 mg q12h for subjects 2 to <6 years of age and ≥ 14 kg, or
  * 150 mg q12h for subjects ≥ 6 years of age.
  Interventions: Drug: Ivacaftor

INTERVENTIONS:
Drug: Ivacaftor
  Other Names: VX-770; Kalydeco
  Arms: Ivacaftor

SUMMARY:
The purpose of this study is to provide information regarding the long-term safety and pharmacodynamics of ivacaftor treatment in the pediatric population younger than 6 years of age with Cystic Fibrosis (CF) who have a CFTR gating mutation in at least 1 allele and will further explore the efficacy of long-term ivacaftor treatment in this population of patients with CF.

ELIGIBILITY:
Inclusion Criteria (Ivacaftor Arm):

1. Completed the last study visit of the treatment period of the previous study (NCT01705145)
2. Hematology, serum chemistry, and vital signs results on Day 1 with no clinically significant abnormalities that would interfere with the study assessments, as judged by the investigator
3. As judged by the investigator, parent or legal guardian must be able to understand protocol requirements, restrictions, and instructions and the parent or legal guardian should be able to ensure that the subject assents to participation in the study to the degree the subject can assent, and that the subject will comply with and is likely to complete the study as planned

Inclusion Criteria (Observational Arm):

1. Subjects who completed their assigned study drug treatment in the previous study (NCT01705145) and elected not to enroll in the ivacaftor arm and subjects who prematurely discontinued treatment in the previous study and received at least 1 dose of study drug treatment in the previous study will be eligible for enrollment in the observational arm.

Exclusion Criteria (Ivacaftor Arm):

1. Subjects who prematurely discontinued from the previous study
2. History of any illness or condition that, in the opinion of the investigator, might confound the results of the study or pose an additional risk in administering study drug to the subject
3. Subjects with a history of study treatment intolerance as observed in their previous study that, in the opinion of the investigator, might pose an additional risk in administering study drug to the subject
4. Subjects receiving commercially-available ivacaftor treatment
5. Subject was unable to complete an adequate slit-lamp examination at the last ophthalmologic examination in the previous study

Exclusion Criteria: (Observational Arm)

1. Subjects receiving ivacaftor treatment will not be eligible for enrollment in the observational arm.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2013-12; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adebayo Lawal, M.D., Study Director — Vertex Pharmaceuticals Incorporated
Locations (16):
- United States (12):
  - Birmingham, Alabama
  - Denver, Colorado
  - Atlanta, Georgia
  - Indianapolis, Indiana
  - Boston, Massachusetts
  - Grand Rapids, Michigan
  - Minneapolis, Minnesota
  - Kansas City, Missouri
  - Omaha, Nebraska
  - Salt Lake City, Utah
  - Richmond, Virginia
  - Seattle, Washington
- Vancouver, British Columbia, Canada
- United Kingdom (3):
  - Edinburgh
  - Liverpool
  - London

REFERENCES:
- [Derived] Rosenfeld M, Cunningham S, Harris WT, Lapey A, Regelmann WE, Sawicki GS, Southern KW, Chilvers M, Higgins M, Tian S, Cooke J, Davies JC; KLIMB study group. An open-label extension study of ivacaftor in children with CF and a CFTR gating mutation initiating treatment at age 2-5 years (KLIMB). J Cyst Fibros. 2019 Nov;18(6):838-843. doi: 10.1016/j.jcf.2019.03.009. Epub 2019 Apr 30. PMID 31053538

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a Phase 3, multicenter, 2 arm study in participants who received at least 1 dose of study drug in parent study VX11-770-108 (study 108) (NCT01705145).
Pre-assignment Details: In study VX11-770-109 (study 109) (NCT01946412), participants were to be enrolled in either ivacaftor arm or observational arm. However, there were no participants enrolled in the observational arm. A total of 33 participants were enrolled in the ivacaftor arm.
Groups:
- Ivacaftor: Participants received ivacaftor 50 milligram (mg) or 75 mg or 150 mg based on body weight and age. Ivacaftor 50 mg administered every 12 hours (q12h) for participants aged 2 to less than (<) 6 years and weighing <14 kilograms (kg), ivacaftor 75 mg q12h for participants aged 2 to <6 years and weighing greater than or equal to (>=) 14 kg and ivacaftor 150 mg q12h for participants >=6 years.
Period: Overall Study
Arm/Group | Ivacaftor
Started | 33
Completed | 28
Not Completed | 5
Not completed — Adverse Event | 1
Not completed — Non-Compliance | 1
Not completed — Continued with commercial Kalydeco | 2
Not completed — Difficulty in swallowing | 1

BASELINE CHARACTERISTICS:
Groups:
- Ivacaftor: Participants received ivacaftor 50 mg or 75 mg or 150 mg based on body weight and age. Ivacaftor 50 mg administered q12h for participants aged 2 to < 6 years and weighing <14 kg, ivacaftor 75 mg q12h for participants aged 2 to <6 years and weighing >= 14 kg and ivacaftor 150 mg q12h for participants >=6 years.
Arm/Group | Ivacaftor
Number analyzed (Participants) | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 3.7 (1.04)
Gender [Count of Participants; unit: Participants]
  Female | 6
  Male | 27

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: AE: any untoward medical occurrence in a participant during the study; the event does not necessarily have a causal relationship with the treatment. This includes any newly occurring event or previous condition that has increased in severity or frequency after the informed consent form is signed. AE includes serious as well as Non-serious AEs. SAE (subset of AE): medical event or condition, which falls into any of the following categories, regardless of its relationship to the study drug: death, life threatening adverse experience, Inpatient hospitalization/prolongation of hospitalization, persistent/significant disability or incapacity, congenital anomaly/birth defect, important medical event. AEs with start date or increased severity on or after the first dose of study drug through the end of study participation was considered treatment-emergent.
Time Frame: Day 1 up to Week 97 (for participants who completed study drug dosing); Day 1 up to 24 weeks after the last dose (up to Week 108, for participants who prematurely discontinued study drug dosing)
Population: Safety set included all participants who received at least 1 dose of study drug in study 109 (NCT01946412). As per the planned analysis for this study, participants were to be analyzed based on their dosing groups as per parent study VX11-770-108 (NCT01705145).
Measure: Number; unit: participants
Groups:
- Ivacaftor 50 mg: Participants who received ivacaftor 50 mg q12h in parent study VX11-770-108 (NCT01705145), received either ivacaftor 50 mg q12h for participants aged 2 to <6 years and weighing <14 kg or ivacaftor 75 mg q12h for participants aged 2 to <6 years and >=14 kg or ivacaftor 150 mg q12h for participants >=6 years in this study (NCT01946412).
- Ivacaftor 75 mg: Participants who received ivacaftor 75 mg q12h in parent study VX11-770-108 (NCT01705145), received either ivacaftor 50 mg q12h for participants aged 2 to <6 years and weighing <14 kg or ivacaftor 75 mg q12h for participants aged 2 to <6 years and >=14 kg or ivacaftor 150 mg q12h for participants >=6 years in this study (NCT01946412).
Arm/Group | Ivacaftor 50 mg | Ivacaftor 75 mg
Number analyzed (Participants) | 9 | 24
participants
  AEs | 9 | 24
  SAEs | 6 | 5

2. Secondary Outcome: Absolute Change From Baseline of Parent Study in Sweat Chloride at Week 24, 48, 72 and 84
Description: Sweat samples were collected using an approved Macroduct (Wescor, Logan, Utah) collection device. A volume of greater than or equal to (>=) 15 microliter was required for determination of sweat chloride. Baseline was defined as the most recent measurement prior to intake of the first dose of study drug in study 108 Part B (NCT01705145).
Time Frame: Baseline (study 108), Week 24, 48, 72 and 84 (study 109)
Population: Safety set. Here "n" signifies those participants who were evaluable at the specified time points for each arm, respectively.As per the planned analysis for this study, participants were to be analyzed based on their dosing groups as per parent study VX11-770-108 (NCT01705145).
Measure: Mean (Standard Deviation); unit: millimole per liter (mmol/L)
Arm/Group | Ivacaftor 50 mg | Ivacaftor 75 mg
Number analyzed (Participants) | 9 | 24
millimole per liter (mmol/L)
  Baseline (n=7,22) | 93.1 (16.2) | 99.6 (13.6)
  Absolute Change at Week 24 (n=6,18) | -62.1 (12.4) | -48.5 (18.4)
  Absolute Change at Week 48 (n=6,15) | -29.3 (37.8) | -51.8 (27.1)
  Absolute Change at Week 72 (n=7,14) | -46.4 (16.0) | -52.9 (26.7)
  Absolute Change at Week 84 (n=6,14) | -46.5 (31.0) | -58.1 (23.9)

3. Secondary Outcome: Absolute Change From Baseline of Study 109 in Sweat Chloride at Week 24, 48, 72 and 84
Description: Sweat samples were collected using an approved Macroduct (Wescor, Logan, Utah) collection device. A volume of >=15 microliter was required for determination of sweat chloride. Baseline is defined as the most recent measurement prior to intake of the first dose of study drug in study 109 (NCT01946412).
Time Frame: Baseline (study 109), Week 24, 48, 72 and 84 (study 109)
Population: Safety set. Here "n" signifies those participants who were evaluable at the specified time points for each arm, respectively. As per the planned analysis for this study, participants were to be analyzed based on their dosing groups as per parent study VX11-770-108 (NCT01705145).
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Ivacaftor 50 mg | Ivacaftor 75 mg
Number analyzed (Participants) | 9 | 24
mmol/L
  Baseline (n= 8,23) | 47.8 (23.3) | 52.9 (23.1)
  Absolute Change at Week 24 (n=7,18) | -4.3 (31.6) | 3.4 (15.9)
  Absolute Change at Week 48 (n=7,17) | 18.1 (39.5) | -4.5 (22.6)
  Absolute Change at Week 72 (n=8,15) | -1.5 (24.3) | -6.0 (20.8)
  Absolute Change at Week 84 (n=7,16) | -2.4 (44.2) | -11.2 (25.4)

4. Secondary Outcome: Absolute Change From Baseline of Parent Study in Weight at Week 12, 24, 36, 48, 60, 72 and 84
Description: Baseline was defined as the most recent measurement prior to intake of the first dose of study drug in study 108 Part B (NCT01705145)
Time Frame: Baseline (study 108), Week 12, 24, 36, 48, 60, 72 and 84 (study 109)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: kilogram (kg)
Arm/Group | Ivacaftor 50 mg | Ivacaftor 75 mg
Number analyzed (Participants) | 09 | 24
kilogram (kg)
  Baseline (n=9, 24) | 12.5 (1.1) | 16.8 (1.8)
  Absolute Change at Week 12 (n= 9, 23) | 1.3 (0.4) | 1.9 (0.7)
  Absolute Change at Week 24 (n=9, 23) | 2.0 (0.6) | 2.5 (0.9)
  Absolute Change at Week 36 (n=9, 23) | 2.4 (0.7) | 3.1 (1.0)
  Absolute Change at Week 48 (n=9, 22) | 2.6 (0.9) | 3.4 (1.1)
  Absolute Change at Week 60 (n=9, 22) | 3.2 (1.0) | 4.0 (1.3)
  Absolute Change at Week 72 (n=9, 20) | 3.4 (0.9) | 4.8 (1.6)
  Absolute Change at Week 84 (n=9, 19) | 4.0 (1.2) | 5.7 (1.9)

5. Secondary Outcome: Absolute Change From Baseline of Study 109 in Weight at Week 12, 24, 36, 48, 60, 72 and 84
Description: Baseline is defined as the most recent measurement prior to intake of the first dose of study drug in study 109 (NCT01946412).
Time Frame: Baseline (study 109), Week 12, 24, 36, 48, 60, 72 and 84 (study 109)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | Ivacaftor 50 mg | Ivacaftor 75 mg
Number analyzed (Participants) | 9 | 24
Kg
  Baseline (n= 9, 24) | 13.5 (1.0) | 18.3 (2.0)
  Absolute Change at Week 12 (n=9, 23) | 0.3 (0.4) | 0.4 (0.5)
  Absolute Change at Week 24 (n=9, 23) | 1.0 (0.5) | 1.0 (0.7)
  Absolute Change at Week 36 (n=9, 23) | 1.4 (0.6) | 1.6 (0.8)
  Absolute Change at Week 48 (n=9, 22) | 1.6 (0.7) | 1.9 (0.8)
  Absolute Change at Week 60 (n=9, 22) | 2.2 (0.8) | 2.5 (1.1)
  Absolute Change at Week 72 (n=9, 20) | 2.4 (0.7) | 3.3 (1.4)
  Absolute Change at Week 84 (n=9, 19) | 3.0 (1.0) | 4.2 (1.7)

6. Secondary Outcome: Absolute Change From Baseline of Parent Study in Stature at Week 12, 24, 36, 48, 60, 72 and 84
Description: Stature was measured as height if children could stand unassisted and follow directions; otherwise, stature was measured as length. Baseline was defined as the most recent measurement prior to intake of the first dose of study drug in study 108 Part B (NCT01705145).
Time Frame: Baseline (study 108), Week 12, 24, 36, 48, 60, 72 and 84 (study 109)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Centimeters (cm)
Arm/Group | Ivacaftor 50 mg | Ivacaftor 75 mg
Number analyzed (Participants) | 9 | 24
Centimeters (cm)
  Baseline (n=9, 24) | 89.1 (4.3) | 102.3 (6.4)
  Absolute Change in Week 12 (n=9, 23) | 4.6 (1.2) | 5.4 (1.1)
  Absolute Change in Week 24 (n=9, 23) | 6.0 (1.7) | 7.7 (3.3)
  Absolute Change in Week 36 (n=9, 23) | 7.8 (1.8) | 8.8 (1.4)
  Absolute Change in Week 48 (n=9, 21) | 9.7 (2.0) | 10.4 (1.7)
  Absolute Change in Week 60 (n=9, 22) | 11.0 (2.2) | 11.6 (2.0)
  Absolute Change in Week 72 (n=9, 20) | 12.5 (2.6) | 13.4 (2.0)
  Absolute Change in Week 84 (n=9, 19) | 13.6 (2.3) | 15.0 (2.3)

7. Secondary Outcome: Absolute Change From Baseline of Study 109 in Stature at Week 12, 24, 36, 48, 60, 72 and 84
Description: Stature was measured as height if children could stand unassisted and follow directions; otherwise, stature was measured as length. Baseline is defined as the most recent measurement prior to intake of the first dose of study drug in study 109 (NCT01946412).
Time Frame: Baseline (study 109), Week 12, 24, 36, 48, 60, 72 and 84 (study 109)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Ivacaftor 50 mg | Ivacaftor 75 mg
Number analyzed (Participants) | 9 | 24
cm
  Baseline (n=9, 24) | 91.7 (4.3) | 105.8 (6.6)
  Absolute Change at Week 12 (n=9, 23) | 2.0 (1.1) | 1.8 (0.9)
  Absolute Change at Week 24 (n=9, 23) | 3.4 (1.2) | 4.1 (3.2)
  Absolute Change at Week 36 (n=9, 23) | 5.2 (1.5) | 5.2 (1.1)
  Absolute Change at Week 48 (n=9, 21) | 7.2 (1.3) | 6.8 (1.3)
  Absolute Change at Week 60 (n=9, 22) | 8.4 (1.4) | 8.0 (1.5)
  Absolute Change at Week 72 (n=9, 20) | 10.0 (2.1) | 9.8 (1.6)
  Absolute Change at Week 84 (n=9, 19) | 11.1 (1.7) | 11.4 (1.9)

8. Secondary Outcome: Absolute Change From Baseline of Parent Study in Body Mass Index (BMI) at Week 12, 24, 36, 48, 60, 72 and 84
Description: BMI = (Weight [in kg]) divided by (Stature [in meters]) ^2. Baseline was defined as the most recent measurement prior to intake of the first dose of study drug in study 108 Part B (NCT01705145).
Time Frame: Baseline (study 108), Week 12, 24, 36, 48, 60, 72 and 84 (study 109)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Kilogram per square meter (kg/m^2)
Arm/Group | Ivacaftor 50 mg | Ivacaftor 75 mg
Number analyzed (Participants) | 9 | 24
Kilogram per square meter (kg/m^2)
  Baseline (n=9, 24) | 15.74 (0.69) | 16.06 (1.15)
  Absolute Change at Week 12 (n=9, 23) | 0.03 (0.40) | 0.09 (0.60)
  Absolute Change at Week 24 (n=9, 23) | 0.31 (0.57) | -0.12 (0.90)
  Absolute Change at Week 36 (n=9, 23) | 0.15 (0.52) | 0.09 (0.73)
  Absolute Change at Week 48 (n=9, 22) | -0.31 (0.60) | -0.13 (0.77)
  Absolute Change at Week 60 (n=9, 22) | -0.12 (0.70) | -0.06 (0.90)
  Absolute Change at Week 72 (n=9, 20) | -0.38 (0.68) | 0.09 (0.97)
  Absolute Change at Week 84 (n=9, 19) | -0.16 (0.96) | 0.28 (0.97)

9. Secondary Outcome: Absolute Change From Baseline of Study 109 in Body Mass Index (BMI) at Week 12, 24, 36, 48, 60, 72 and 84
Description: BMI = (Weight [in kg]) divided by (Stature [in meters]) ^2. Baseline is defined as the most recent measurement prior to intake of the first dose of study drug in study 109 (NCT01946412).
Time Frame: Baseline (study 109), Week 12, 24, 36, 48, 60, 72 and 84 (study 109)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Ivacaftor 50 mg | Ivacaftor 75 mg
Number analyzed (Participants) | 9 | 24
kg/m^2
  Baseline (n= 9, 24) | 16.07 (0.55) | 16.33 (1.12)
  Absolute Change at Week 12 (n= 9, 23) | -0.30 (0.60) | -0.16 (0.48)
  Absolute Change at Week 24 (n= 9, 23) | -0.02 (0.70) | -0.36 (1.03)
  Absolute Change at Week 36 (n= 9, 23) | -0.18 (0.83) | -0.16 (0.63)
  Absolute Change at Week 48 (n= 9, 22) | -0.64 (0.81) | -0.35 (0.57)
  Absolute Change at Week 60 (n= 9, 22) | -0.45 (0.82) | -0.29 (0.72)
  Absolute Change at Week 72 (n= 9, 20) | -0.71 (0.90) | -0.21 (0.78)
  Absolute Change at Week 84 (n= 9, 19) | -0.49 (1.09) | -0.01 (0.87)

ADVERSE EVENTS:
Time Frame: Day 1 up to Week 97 (for participants who completed study drug dosing); Day 1 up to 24 weeks after the last dose (up to Week 108, for participants who prematurely discontinued study drug dosing)
Description: As per the planned analysis for this study, participants were to be reported based on their dosing groups as per parent study VX11-770-108 (NCT01705145).
Arm/Group | Ivacaftor 50 mg | Ivacaftor 75 mg
Serious Adverse Events (participants affected / at risk) | 6/9 | 5/24
Other Adverse Events (participants affected / at risk) | 9/9 | 24/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ivacaftor 50 mg (N=9) | Ivacaftor 75 mg (N=24)
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 3 | 3
Enterovirus infection (Infections and infestations) | 0 | 1
Respiratory syncytial virus infection (Infections and infestations) | 1 | 0
Staphylococcal infection (Infections and infestations) | 0 | 1
Alanine aminotransferase increased (Investigations) | 2 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 0
Adenovirus test positive (Investigations) | 1 | 0
Pyrexia (General disorders) | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Seizure anoxic (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ivacaftor 50 mg (N=9) | Ivacaftor 75 mg (N=24)
Otitis media (Infections and infestations) | 2 | 4
Sinusitis (Infections and infestations) | 2 | 3
Viral upper respiratory tract infection (Infections and infestations) | 0 | 5
Gastroenteritis viral (Infections and infestations) | 0 | 4
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 0 | 4
Pharyngitis streptococcal (Infections and infestations) | 1 | 3
Nasopharyngitis (Infections and infestations) | 1 | 2
Rhinitis (Infections and infestations) | 2 | 1
Bronchitis (Infections and infestations) | 1 | 1
Respiratory tract infection viral (Infections and infestations) | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 1 | 1
Varicella (Infections and infestations) | 0 | 2
Ear infection (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Hand-foot-and-mouth disease (Infections and infestations) | 0 | 1
Herpangina (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 0 | 1
Lower respiratory tract infection bacterial (Infections and infestations) | 0 | 1
Lung infection pseudomonal (Infections and infestations) | 0 | 1
Molluscum contagiosum (Infections and infestations) | 0 | 1
Myringitis (Infections and infestations) | 0 | 1
Parainfluenzae virus infection (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Rhinovirus infection (Infections and infestations) | 0 | 1
Staphylococcal skin infection (Infections and infestations) | 0 | 1
Streptococcal infection (Infections and infestations) | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 1
Upper respiratory tract infection bacterial (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 16
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Allergic sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiration abnormal (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Snoring (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 6 | 7
Abdominal pain (Gastrointestinal disorders) | 0 | 5
Constipation (Gastrointestinal disorders) | 1 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 0
Tooth discolouration (Gastrointestinal disorders) | 0 | 1
Pyrexia (General disorders) | 7 | 6
Fatigue (General disorders) | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 4
Aspartate aminotransferase increased (Investigations) | 1 | 3
Bacterial test positive (Investigations) | 1 | 1
Gamma-glutamyltransferase increased (Investigations) | 1 | 1
Haemophilus test positive (Investigations) | 0 | 2
Respiratory rate increased (Investigations) | 1 | 1
Adenovirus test positive (Investigations) | 1 | 0
Antibiotic resistant Staphylococcus test positive (Investigations) | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 1
Influenza A virus test positive (Investigations) | 0 | 1
Lymph node palpable (Investigations) | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 1
Pseudomonas test positive (Investigations) | 1 | 0
Respiratory syncytial virus test positive (Investigations) | 1 | 0
Staphylococcus test positive (Investigations) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 3 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 1
Red man syndrome (Skin and subcutaneous tissue disorders) | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 1 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Eye injury (Injury, poisoning and procedural complications) | 0 | 1
Conjunctivitis (Eye disorders) | 2 | 0
Amblyopia (Eye disorders) | 0 | 1
Cataract cortical (Eye disorders) | 0 | 1
Eye pruritus (Eye disorders) | 0 | 1
Lacrimation increased (Eye disorders) | 0 | 1
Ear pain (Ear and labyrinth disorders) | 1 | 1
Cerumen impaction (Ear and labyrinth disorders) | 0 | 1
Convulsion (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Lethargy (Nervous system disorders) | 1 | 0
Migraine (Nervous system disorders) | 0 | 1
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 0 | 1
Encopresis (Psychiatric disorders) | 0 | 1
Onychophagia (Psychiatric disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Enuresis (Renal and urinary disorders) | 0 | 1
Micturition urgency (Renal and urinary disorders) | 1 | 0
Phimosis (Congenital, familial and genetic disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI is free to publish results of the study after (1) the first multi-center publication, (2) if the sponsor elects not to publish the results, or (3) 18 months after close of the study, whichever occurs first. Proposed publications are to be submitted to the sponsor for review and comment for a period of at least 45 days (which may be extended under certain circumstances related to protection of intellectual property); the sponsor cannot require changes to the proposed publications.